CLINICAL TRIAL: NCT04821908
Title: Consequences of SARS-CoV2 Pandemic on Childhood Asthma Control and Exacerbations: French Multicenter Cross-sectional VIRASTHMA COVID G4 Study
Brief Title: Consequences of COVID 19 Pandemic on Childhood Asthma
Acronym: VIRASTHCOVID
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2020_85; 2020-A03365-34 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2021-03-29; First posted 2021-03-30 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-12

CONDITIONS: Asthma in Children
Keywords: Asthma control; COVID-19 pandemic; Respiratory infection; Environmental pollution
MeSH Terms: conditions — COVID-19; Respiratory Tract Infections

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — plasma nasal swab
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: population included in the VIRASTHMA COVID G4 study
- Group 2: population included in the previous studies "VIRASTHMA", "CHAMPIASTHMA" (IRDCB No.: 2019-A03310-57), "COBRAPED" (NCT02114034), "VIRASTHMA 2" (IRDCB No.: 2014 A01687 40, NCT: 03960359), "INCOVPED" (pediatric emergencies, NCT04336761).

SUMMARY:
The SARS-CoV2 pandemic, which emerged in the first quarter of 2020, has led to an unprecedented health crisis in our modern healthcare systems and has resulted in strong national public health measures. The impact of the pandemic and its indirect environmental consequences on pediatric asthma is currently being assessed. In particular, the study of its role on the risk of exacerbations and modification of control is one of the priority research objectives defined by European societies.

The primary aim is to study the impact of the pandemic on asthma control in children aged 3-16 years with a medical diagnosis of asthma, compared to data from other observational cohorts conducted in the same region prior to the pandemic.

A sub-population of children 3-16 years will be assessed at exacerbation and at a follow-up visit, 2-4 months later, with clinical data, biological and microbiological samples.

DETAILED DESCRIPTION:
Children aged 3-16 years with a medical diagnosis of asthma, will be assessed for asthma control, exacerbation rate.

Data will be compared to data from other observational cohorts conducted in the same region prior to the pandemic.

A sub-population of children 3-16 years will be assessed at exacerbation and at a follow-up visit, 2-4 months later, with clinical data, biological and microbiological samples.

ELIGIBILITY:
Inclusion Criteria:

* Children and adolescents aged 3 to 16 years old
* With a medical diagnosis of asthma as per-guidelines, who had been followed-up for at least 6 months,
* Assessed in one of the pediatric departments participating in the study,
* After written consent of at least one of the 2 parents and/or representative of the parental authority, and of the child if he is older than 8 years old.

Criteria for the sub-population assessed at "exacerbation" and second visit:

* Children and adolescents aged 3 to 16 years
* With a medical diagnosis of asthma as per-guidelines, who had been followed-up for at least 6 months,
* Hospitalized for a severe asthma exacerbation (requiring hospitalization and general corticosteroid therapy) at Lille University Hospital
* After written consent of both parents and/or representative of the parental authority, and of the child if he is over 8 years old

Exclusion Criteria:

* History of chronic respiratory disease other than asthma,
* Inability of parents to receive informed information, inability to participate in the entire study, refusal to sign the consent form

Ages: 3 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: children and adolescents diagnosed with asthma.
Sampling Method: Probability Sample
Enrollment: 577 (Estimated)
Dates: Start 2021-09-14 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Controlled asthma | at inclusion
  Composite criteria defined by a cACT (4-11 years) or ACT (12-16 years) score ≥ 20 and according to GINA criteria.

SECONDARY OUTCOMES:
Characteristics of asthma | At inclusion and follow-up visit at 2-4 months for the sub-population included at exacerbation
  Composite criteria : allergic phenotype, severity assessed by GINA treatment level, number of exacerbations in the past year, lung function
history of SARS-Cov2 infection in the past year | At inclusion and Follow-up visit at 2-4 months for the sub-population included at exacerbation
  history of SARS-Cov2 infection based on patient report
number of infectious episodes in the past year | At inclusion and Follow-up visit at 2-4 months for the sub-population included at exacerbation
  number of infectious episodes based on patient report
Observance | At Inclusion and Follow-up visit at 2-4 months for the sub-population included at exacerbation
  Assessed by four-items Morisky-Green questionnaire : 1/ Do you ever forget to take your medication; 2/ Are you careless sometimes about taking your medication 3/ When you feel better, do you sometimes stop taking your medication 4/ Sometimes, if you feel worse when you take your medication, do you stop taking it. An answer "no" to any of the 4 questions is considered as "not well-observed medication".
QoL (Quality of life) in children aged 7-17 years | At Inclusion and Follow-up visit at 2-4 months for the sub-population included at exacerbation
  Assessed by PAQLQ : PAEDIATRIC ASTHMA QUALITY OF LIFE QUESTIONNAIRE. The PAQLQ has 23 questions in 3 domains (symptoms, activity limitation and emotional function). The activity domain contains 3 'patient-specific' questions. Children are asked to think about how they have been during the previous week and to respond to each of the 32 questions on a 7-point scale (7 = not bothered at all -
  1 = extremely bothered). The overall PAQLQ score is the mean of all 23 responses and the individual domain scores are the means of the items in those domains. The highest the score is, the better QoL is.
Outdoor levels of pollutants and pollens | At Inclusion and Follow-up visit at 2-4 months for the sub-population included at exacerbation
  Composite criteria : monthly average measurements of CO, O3, NO, NO2, SO2, PM2.5, PM10 and pollen counts
Respiratory virus infection (SARS-CoV2 and other) | at exacerbation and at follow-up visit at 2-4 months for the sub-population included at exacerbation
  Results of viral PCR

CONTACTS AND LOCATIONS:
Overall Officials: Stéphanie Lejeune, MD, Principal Investigator — University Hospital, Lille
Locations (1):
- CHU Lille, Lille, France